CLINICAL TRIAL: NCT03130192
Title: An Observational Study of the Correlation Between Cancer-related Fatigue, Survival and Physiological Factors in Non-Small Cell Lung Cancer (NSCLC) Patients Under Chemotherapy
Brief Title: A Study of the Correlation Between CRF, Survival and Physiological Factors in NSCLC Patients Under Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, LJ Hwu, Institutional review board, Chung Shan Medical University
Other Study IDs: CSMUH01
Record Dates: First submitted 2017-03-26; First posted 2017-04-26 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Worldwide, non-small cell lung cancer (NSCLC) is one of the most common causes of cancer mortality. Also, the first leading cause of death is lung cancer in Taiwan 2012. Most patients are diagnosed at advanced stages and their median survival with supportive care is only 3-6 months. The common regimens used on advanced NSCLC treatment consists of platinum-based doublet chemotherapy, the survival benefit of which is able to extend the survival to approximately 10 months. However, disease and treatment-related toxicities in cancer patients may result in fatigue and interfered quality of life (QoL). According to the others reports, eight QoL areas including physical functioning, fatigue, pain, and appetite loss have been showed a statistically significant association with survival rate of NSCLC patients.

Cancer-related fatigue (CRF), an indicator of QoL, has been reported as the most frequent and distressing toxicity of lung cancer chemotherapy. Proposed criteria for CRF have been adopted for inclusion in the International Statistical Classification of Disease and Related Health Problems, Tenth Revision, Clinical Modification (ICD-10-CM). Therefore, more in-depth researches on CRF are needed in Taiwan.

In addition, electrolyte disturbance like hyponatremia has been reported to be counted as one of the many contributing factors for fatigue in palliative care patients and associated with poorer overall survival rate (OS) in lung cancer. Thus, the correlation between CRF and electrolyte possibly would be a strong link for physician to improve the QoL and survival rate of NSCLC patients.

The objective of this observational study is to evaluate the correlation between CRF, survival and physiological factors in NSCLC patients under chemotherapy. The study will compare the effect of QoL and CRF on survival with or without CRF treatment and investigate the correlation between the variation of CRF and physiological factors which have been examined and recorded on medical record under clinical practice. These results will supply physicians with more understanding about CRF, and help them to enhance the quality on lung cancer care to being perfected in the future.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) patients with chemotherapy will be enrolled. Patients will be thoroughly informed about all aspects of the study activity schedule and all regulatory requirements that must be satisfied for informed consent. Only patients who give consent to participate in this study and meet all other inclusion and exclusion criteria will be eligible to enroll into this study. ICD-10 fatigue criteria, Brief Fatigue Inventory-Taiwan Form (BFI-T), the visual analog scale (VAS) for appetite and Functional Assessment of Cancer Therapy-General quality of life questionnaire (FACT-G7) will be used to evaluate patients' fatigue and quality of life. Patients who enrolled in this observational study will complete the evaluation and questionnaire of fatigue and quality of life according to clinical schedule. The first survey (baseline) will be collected after enrollment, the further surveys will be completed every three chemotherapy cycles following subject's chemotherapy schedule and after finish the whole course of chemotherapy. Subject demographic and disease-related information and routine laboratory data will also be collected from medical record for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who signed the informed consent form.
* Aged 20 years and older.
* Patients who have been given a diagnosis of stage II-IV NSCLC cancer.
* Patients who are under/ or scheduled for chemotherapy treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Patients who are able to complete QoL questionnaires.

Exclusion Criteria:

* Patients have enrolled or have not yet completed other investigational drug trials within 30 days before screening.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer (NSCLC) patients with chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-12-22 (Actual); Primary Completion 2021-06-07 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Cancer-related fatigue evaluation by brief fatigue inventory-Taiwanese form (BFI-T) | Change from baseline cancer-related fatigue at 6 chemotherapy cycles (24 weeks)

SECONDARY OUTCOMES:
Quality of life assessments by functional assessment of cancer therapy-general 7 (FACT-G7) | Change from baseline quality of life at 6 chemotherapy cycles (24 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No